CLINICAL TRIAL: NCT01204359
Title: "5010 Clinical Research Programme"of Sun Yat-sen University
Brief Title: The Prospective Study of Standard Treatment of Graves Disease Iodine 131 and Prevention of Adverse Reactions
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: ningyi jiang, SUN YAT-SEN UNIVERSITY
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2007022
Record Dates: First submitted 2010-09-15; First posted 2010-09-17 (Estimated); Last update posted 2015-05-25 (Estimated); Status verified 2015-05

CONDITIONS: Hypothyroidism; Exophthalmos
MeSH Terms: conditions — Hypothyroidism; Exophthalmos | interventions — Iodine-131

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- follow-up (No Intervention)
  Interventions: Radiation: Iodine 131

INTERVENTIONS:
Radiation: Iodine 131 — iodine 131，185、370、555mBq，6 months

SUMMARY:
Iodine 131 (131I） treatment on Graves disease and Graves ophthalmopathy relationship has always been the focus of debate. Majority view is that the current treatment does not increase 131I Graves ophthalmopathy, therefore,Graves disease associated with exophthalmos is not a contraindication of 131I treatment. While treatment with corticosteroids, a timely corrective measures to be effective in preventing Graves ophthalmopathy adverse effects. But the merger with severe proptosis in patients with Graves , especially infiltrative exophthalmos , the application of 131I treatment will induce or aggravate not yet reached consensus, so, the 131I treatment is still very careful , mainly due to plaque prospective study and visual assessment is not lack of uniform standards, and a variety of factors (including smoking, work status, and 131I treatment of thyroid doses, etc.) may also interfere or influence the ultimate effect of 131I on the Graves ophthalmopathy. In the view of this situation Graves disease patients with Graves ophthalmopathy could be 131I treatment or not, how to dose adjustments, and the use of which required treatment with systemic issues such as research, explore treatment exophthalmos reduction and mitigation of increased proptosis reasonable treatment of symptoms. To further promote the standardization of 131I treatment of Graves disease on basis.

DETAILED DESCRIPTION:
no more description

ELIGIBILITY:
Inclusion Criteria:

* a typical clinical symptoms of Graves disease, diffuse goiter, eye signs (including exophthalmos), thyroid function (FT3, FT4, rTSH) and thyroid autoantibodies and imaging examinations to confirmed.

Exclusion Criteria:

* 131I treatment contraindications, those who have not signed the informed consent, failure to complete treatment and follow-up estimates of patients and patients not suitable for radionuclide therapy

Ages: 8 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 627 (Estimated)
Dates: Start 2007-07; Primary Completion 2016-07 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
The rate of Hypothyroidism after Iodine 131 treatment | one year

SECONDARY OUTCOMES:
The side effect to Infiltrative exophthalmos after Iodine 131 treatment | one year

CONTACTS AND LOCATIONS:
Overall Officials: SUN YAT-SEN UNIVERSITY ningyi jiang, professor, Principal Investigator — Sun Yat-sen University
Locations (2):
- China (2):
  - Sun Yat-sen Memorial Hospital, Guangzhou, Guangdong
  - Ningyi Jiang, Guangzhou